CLINICAL TRIAL: NCT05171374
Title: Prospective Evaluation of Clinical Outcomes in Patients With Resectable or Metastatic BRAF+ Melanoma Treated With Dabrafenib and Trametinib in Real Practice
Brief Title: pRospective Evaluation of Clinical Outcomes in Patients With metAsTatIс melanOma Treated With dabrafeNib and trAmetinib in reaL practicE
Acronym: RATIONALE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MelanomaPRO, Russia (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CDRB436ARU01R / MELPRO-0721
Record Dates: First submitted 2021-09-27; First posted 2021-12-28 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; Melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adjuvant cohort: Patients with resectable stage III melanoma, reciveng dabrafenib and trametinib in adjuvant settings
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Metastatic cohort: Patients with unresectable stage IIIC/D or stage IV melanoma, reciveng dabrafenib and trametinib in metastatic settings
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Observational stusy. No intervention is planned
Drug: Trametinib — Observational stusy. No intervention is planned

SUMMARY:
Prospective evaluation of clinical outcomes in patients with resectable or metastatic BRAF+ melanoma treated with dabrafenib and trametinib in real practice

DETAILED DESCRIPTION:
Rationale and background It is now accepted by the majority of experts in oncology that most effective and safe therapy options should be considered for first-line treatment, including adjuvant setting. As the routine administration of drugs including dosing, treatment interruptions, and early termination in clinical practice may vary from procedures used in clinical trials, post-authorization "real-world" data are important to quantify feasibility, acceptance, and practical considerations on prescription of targeted therapy with Dabrafenib+Trametinib. Therefore, it is of great interest for clinical and scientific communities to evaluate patient and treatment choice used in routine practice of Russian oncology centers. The aim of this study is to asses clinical outcomes of patient receiving Dab+Tram in different substages of resectable melanoma and different lines in metastatic melanoma., Additionally, it is of interest to gain insights into real world data regarding quality of life of melanoma patients treated with Dabrafenib and Trametinib in adjuvant or metastatic setting.

Research question and objectives Primary objective The primary objective in the study is to estimate relapse-free survival (RFS) in melanoma patients in adjuvant settings and progression free survival (PFS) in melanoma patients in metastatic settings. Primary endpoints

• The primary efficacy endpoint of the study is 12-month RFS rate, definded as the time form index date to the date of first documented relapse or death due to any cause.

The primary efficacy endpoint of the study is 12-month PFS rate, defined as the time from the index date to the date of the first documented progression by investigator judgement or death due to any cause. If a patient has not had an event, PFS will be censored at the date of the last tumor assessment

Secondary objectives

* To describe patient populations receiving dabrafenib and trametinib for stage III resectable melanoma with respect to demographics and clinical characteristics at index date (baseline).
* To describe patient populations receiving dabrafenib and trametinib for stage IV metastatic melanoma with respect to demographics and clinical characteristics at index date (baseline).
* Evaluate retrospectively the sequence of therapy prior to initiating treatment with Dabrafenib and Trametinib.
* Analyze prospectively treatment options following disease recurrence or progression on treatment with Dabrafenib and Trametinib.
* Analyze proportion (%) of patients receiving adjuvant therapy with Dabrafenib and Trametinib for melanoma stage IIIA/IIIB/IIIC/IIID
* Analyze proportion (%) of patients receiving Dabrafenib and Trametinib in 1L/2L/3L/later lines in metastatic settings.
* Assess clinical outcomes (including treatment duration, treatment discontinuation rate) in melanoma patients treated with Dabrafenib and Trametinib in adjuvant settings in real-world practice.
* Assess clinical outcomes in melanoma patients treated with Dabrafenib and Trametinib in metastatic settings (including median PFS, treatment duration, RR and) in real-world practice.
* Assess safety of therapy of interest: rate of adverse events associated with the therapy, proportions of patients and reasons of dose adjustment on dabrafenib and trametinib, discontinuation rate and reasons of discontinuation in melanoma patients treated with Dabrafenib and Trametinib in adjuvant and metastatic in real-world practice.
* Describe changes in patient-reported symptoms and quality of life (QoL) in melanoma patients treated with Dabrafenib and Trametinib in real-world setting.

Study design Patients will attend study sites in accordance with routine clinical practice. It is assumed that visits will performed every 3-4 months, as it is stated by the current guidelines (1). Patients will undergo standard procedures and tests according to clinical guidelines and physician's judgement (1). Available data from routine clinical management of the patients will be collected in the course of visits to investigation site.

The supposed duration of observation within the study is 1 year which corresponds to the requested duration of adjuvant therapy and is in line with the median PFS - 11.1 months according to the COMBI D/V trials' analysis for dabrafenib+trametinib therapy in the first line treatment of metastatic cutaneous melanoma with BRAF mutation (2). The enrollment period will continue for two years.

Baseline assessments will include collection of patient demographic data, disease history, treatment history, laboratory data and physical examination results as assessed by clinicians and patient reported outcomes (PROs) for symptoms and QoL. Treatment history will include all pharmacological therapy, its duration, response duration, reason for discontinuation. QoL assessment is not a part of routine practice for some investigation sites, hence, QoL will be evaluated if it does not interfere routine practice.

At each following visit (as indicated above, approximately each 3-4 months up to 1 year) available information on treatment status, response and progression, PROs, patient performance status and any relevant adverse occurrences will be collected.

Setting and study population This study is planned as a prospective non-interventional multicenter study. This study is observational in nature and does not impose a therapy protocol, diagnostic/therapeutic interventions or a visit schedule. Patients with resectable or metastatic BRAF+ melanoma, in that treatment with dabrafenib and trametinib was initiated, either newly diagnosed or progressive during prior lines of therapy, will be included into the study. Initiation of dabrafenib+trametinib therapy will be considered an index event.

Adult patients receiving dabrafenib and trametitnib for adjuvant or metastatic melanoma treatment will be enrolled into study.

Variables All data will be collected in the course of prospective visits of patient to the clinical site according to routine practice. Demographic, disease and treatment-related variables will be collected in order to ensure completeness of data for endpoint analysis. Definitions of variables for analysis will be given in the relevant section of protocol.

Data sources Medical records and other disease-related documents will be used in the study.

Study size This study does not test any pre-defined statistical hypotheses therefore sample size and power calculation projections are not applicable. Since there is no formal hypothesis-testing, sample size for this study is based on the feasibility of enrolling the desired population during the enrolment period for this study.

Data analysis This is an exploratory study and no comparative analysis is planned. Descriptive statistics will be tabulated for the demographic and clinical characteristics and outcome variables. In all cases, point estimates as well as the corresponding two-sided 95% CI will be presented. No missing value imputation will be performed.

Kaplan-Meier method will be used for the analysis of time-to-event.

Milestones

Planned dates of study milestones:

Concept approved: 29 April 2021 Final protocol approval: 30 June 2021 Start of data collection (FPFV): 30 September 2021 End of enrollment (LPFV): 30 September 2023 End of primary data collection (LPLV): 30 September 2024 Final report on study results: 30 April 2025 Publication of study results: 30 September 2025

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older;
* Histologically confirmed stage III resectable or stage IV metastatic cutaneous melanoma with confirmed BRAF mutation, for whom the treating physician took the decision to initiate treatment with dabrafenib and trametinib before entering the study;
* Treatment with Dabrafenib and Trametinib was initiated no longer than 4 weeks (28 days) prior to written informed consent for this study;
* Performance status ≤ 2 by Eastern Cooperative Oncology Group (ECOG) scale;
* Patient is willing and able to participate in the study;
* Written informed consent for study participation.

Exclusion Criteria:

* Patients with a life expectancy of less than 3 months at the time of melanoma diagnosis, per the investigator's judgment.
* Patients participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment. (Patients participating in other investigator initiated or other non-interventional study [NIS] can be included as long as their standard of care is not altered by the study).
* Patients on active treatment for malignancies other than melanoma at the time of enrollment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study will be conducted in investigation sites specialized in treatment of solid neoplasm or, more narrowed, melanoma. Patient may be enrolled either by surgical or medical oncologist if relevant indormation is available and there is no obvious risk for loss of contact with patient. Study population will be formed of the patients from cancer treatment facilities and the representativeness of sample may vary depending on participating sites. Study is going ro include patients receiving treatment of interest (dabrafenib and trametinib) for either adjuvant of metastatic setting of melanoma treatment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
12-month RFS rate | 12 months
  The primary efficacy endpoint of the study is 12-month RFS rate, definded as the time form index date to the date of first documented relapse or death due to any cause
12-month PFS rate | 12 months
  The primary efficacy endpoint of the study is 12-month PFS rate, defined as the time from the index date to the date of the first documented progression by investigator judgement or death due to any cause. If a patient has not had an event, PFS will be censored at the date of the last tumor assessment

SECONDARY OUTCOMES:
To describe patient populations receiving dabrafenib and trametinib for stage III resectable melanoma with respect to demographics and clinical characteristics at index date (baseline). | 12 months
To describe patient populations receiving dabrafenib and trametinib for stage IV metastatic melanoma with respect to demographics and clinical characteristics at index date (baseline) | 12 months
Evaluate retrospectively the sequence of therapy prior to initiating treatment with Dabrafenib and Trametinib | 12 months
Analyze prospectively treatment options following disease recurrence or progression on treatment with Dabrafenib and Trametinib | 12 months
Analyze proportion (%) of patients receiving adjuvant therapy with Dabrafenib and Trametinib for melanoma stage IIIA/IIIB/IIIC/IIID | 12 months
Analyze proportion (%) of patients receiving Dabrafenib and Trametinib in 1L/2L/3L/later lines in metastatic settings | 12 months
To assess treatment duration in melanoma patients treated with Dabrafenib and Trametinib in adjuvant settings in real-world practice | 12 months
To assess treatment discontinuation rat in melanoma patients treated with Dabrafenib and Trametinib in adjuvant settings in real-world practice | 12 months
To assess median PFS in melanoma patients treated with Dabrafenib and Trametinib in metastatic settings in real-world practice | 12 months
To assess median treatment duration in melanoma patients treated with Dabrafenib and Trametinib in metastatic settings in real-world practice | 12 months
To assess treatment discontinuation rate in melanoma patients treated with Dabrafenib and Trametinib in metastatic settings in real-world practice | 12 months
To assess rate of adverse events associated with the therapy of interest | 12 months
To assess proportions of patients and reasons of dose adjustment on dabrafenib and trametinib in melanoma patients treated with Dabrafenib and Trametinib in adjuvant and metastatic in real-world practice | 12 months
Description of changes in patient-reported symptoms and quality of life (QoL) in melanoma patients treated with Dabrafenib and Trametinib in real-world setting | 12 months

CONTACTS AND LOCATIONS:
Locations (15):
- Russia (15):
  - Altai Regional Oncological Dispensary, Barnaul, Alatai
  - Republican Clinical Oncology Center of Chuvashia, Cheboksary, Chuvashskaya Respublika
  - Irkutsk Regional Oncological Dispensary, Irkutsk, Irkutsk Oblast
  - Rostov Regional Oncological Dispensary, Rostov-on-Don, Rostov Oblast
  - State Budget Health Institution of the Republic of Mordovia "Republican Oncological Dispensary", Saransk, THE Republic of Mordovia
  - Republican Clinical Oncological Dispensary named after Sergei Grigoryevich Primushko Ministry of Health of the Udmurt Republic, Izhevsk, The Udmurt Republic
  - Ivanovo Regional Oncological Dispensary, Ivanovo
  - KGBUZ "Krasnoyarsk regional clinical oncological dispensary named after A.I. A.I. Kryzhanovsky", Krasnoyarsk
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - Moscow City Clinical Oncology Hospital No. 1, Moscow
  - Omsk Regional Clinical Oncology Center, Omsk
  - Perm Regional Oncological Dispensary, Perm
  - Tambov Regional Oncological Clinical Dispensary, Tambov
  - Sverdlovsk Regional Oncology Center, Yekaterinburg
  - GBUZ Yuzhno-Sakhalinsk oncologic dispensary, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: No